CLINICAL TRIAL: NCT04778098
Title: The Use of an SMS Reminder in Postoperative Medication Compliance in Patients Undergoing Cataract Surgery and Its Effect on Anxiety: A Randomized Controlled Study
Brief Title: Effect of Short Message Service Use on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Figen Dıgın, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/P0244
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Cataract
Keywords: anxiety; satisfaction; surgery; telenursing; text message
MeSH Terms: conditions — Cataract; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS group (Experimental): After postoperative standard discharge education was provided to the patients in the SMS group, they were given an individualized written Postoperative Medication Reference Chart. The patient/relative, whose contact information was received, was informed that they would be reminded via text message (SMS). SMS reminders which were individualized according to the patient based on the doctor's directive, were sent to the patients in the SMS group by the researcher clinical nurse (A. Ş). SMS sending started on postoperative day 1 and ended on day seven.
  SAI was applied again to all patients who came to the outpatient clinic for control on postoperative day seven. Unlike the control group, the "Patient Satisfaction Form," which was prepared for the use of SMS reminders, was applied to the patients in the SMS group. Confirmation was obtained from the patients and their relatives that SMS reminders were received every day.
  Interventions: Other: Received SMS reminder
- Control group (No Intervention): the Patient Identification Form and SAI were applied to patients in the control on the day of surgery (postoperative day 0). Routine discharge education was provided to all patients by clinical nurses. During the discharge of the patients in the control group, they were informed about the change of dressing on the next day (postoperative day one) and control in the outpatient clinic on postoperative day seven. The patients were given an individualized written Postoperative Medication Reference Chart indicating the dosage and application time of eye drops they must follow for seven days at home.

INTERVENTIONS:
Other: Received SMS reminder — telenursing
  Arms: SMS group

SUMMARY:
Background: Paticipants undergoing cataract surgery find postoperative medication management difficult and are anxious about this issue. Differences in the number of medications and frequency of administration can be lead to confusion in participants.

Aims and objectives: The aim of this randomized-controlled study was to evaluate the effect of using SMS, which reminds about the intake of medication, on reducing postoperative anxiety in participants undergoing cataract surgery.

Design: Randomized controlled study.

DETAILED DESCRIPTION:
This randomized controlled study was conducted with the participation of 82 patients in the ophthalmology clinic of a private hospital between July 2020 and February 2021. Participants who underwent cataract surgery in a private hospital constituted the population of the study. Based on the findings in the literature (Karaman Özlü et al., 2016) (mean score of the State Anxiety Inventory 27.54±3.25), the minimum number of participants to be included in the sample was determined to be 82 (41 subjects-41 controls), each group consisting of 41 people by predicting a confidence interval of 99.9%, an error rate of 5%, and a power of 95%.

Participants who were adults, volunteered to participate in the study, accepted randomization, could communicate in Turkish, had a personal cell phone, could read text messages or were illiterate and had a relative to help participants at home after discharge were included in the study.

Data Collection Tools The study data were collected using the Patient Identification Form and Patient Satisfaction Form.

Patient Identification Form: The form prepared by the investigater with the help of the literature (Gülşen & Akansel, 2020; & Lim et al., 2018) consisted of 8 questions examining the individual variables (age, gender, education level, marital status, comorbidity, working status and the patient's state of living alone, and the experience of cataract).

State Anxiety Inventory (SAI) In 1970, Spielberg et al. developed the State Anxiety Inventory, and Oner and Le Compte carried out its reliability and validity studies. According to 20 expressions with inventory, the individual may determine his or her feelings at a specific location and time. The State Anxiety Inventory are scored between 20 and 80. A higher score suggests a high anxiety level. The Cronbach alpha for Turkish version of the SAI was 0.94 to 0.96 (Öner & Le Compte, 1983; Öner, 2008). In this study, the coefficient of Cronbach alpha was calculated to be 0.93 for the inventory.

Patient Satisfaction Form The form consisted of one question about participants' satisfaction with receiving an SMS reminder. The satisfaction level of participants was classified into four levels. The value "0" was determined as "Not satisfied at all," and the value "3" was determined as "Very satisfied." Postoperative Medication Reference Chart It is a "chart" including the dosage and application time of all eye drops until postoperative day seven, which is the second control of the participant according to the doctor's directive. Medications were individualized for each participant by the investigater clinical nurse according to the doctor's directive.

Data Collection Before starting the data collection, 82 participants who met the sampling acceptance criteria were prospectively identified.

The investigater provided information about the study, the aim and significance of the study, and the investigater to the individuals hospitalized in the ophthalmology service for cataract surgery, and then informed consent was obtained in writing from the individuals. Randomization was done by coin tossing (those who came up tails were included in the SMS group, and those who came up heads were included in the control group), and according to the results, the Patient Identification Form and SAI were applied to all participants in the control and SMS groups on the day of surgery (postoperative day 0). Routine discharge education was provided to all participants by clinical nurses. During the discharge of the participants in the control group, they were informed about the change of dressing on the next day (postoperative day one) and control in the outpatient clinic on postoperative day seven. The participants were given an individualized written Postoperative Medication Reference Chart indicating the dosage and application time of eye drops participants must follow for seven days at home.

SMS group After postoperative standard discharge education was provided to the participants in the SMS group, participants were given an individualized written Postoperative Medication Reference Chart indicating the dosage and application time of eye drops participants must follow for seven days at home. The participants/relative, whose contact information was received, was informed that they would be reminded via SMS. SMS reminders such as "Dear x, do not forget to apply your eye drop called X as 5 drops three times a day and your eye drop called X as 2 drops three times a day. Investigater hope you get well soon," which were individualized according to the participant based on the doctor's directive, were sent to the participants in the SMS group by the investigater clinical nurse (A. Ş). SMS sending started on postoperative day 1 and ended on day seven.

SAI was applied again to all participants who came to the outpatient clinic for control on postoperative day seven. Unlike the control group, the "Patient Satisfaction Form," which was prepared for the use of SMS reminders, was applied to the participants in the SMS group. Confirmation was obtained from the participants and their relatives that SMS reminders were received every day.

Randomization Randomization (1:1 allocation ratio) was determined by the simple randomization method (coin tossing). As a result of coin tossing, participants who came up tails were allocated to the SMS group (n = 41), and participants who came up heads were allocated to the control group (n = 41), (Figure 1).

Blinded Due to the nature of the intervention, the participants and the investigaters could not be blinded to the intervention (SMS sending) since open participation was required.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were adults, volunteered to participate in the study, accepted randomization, could communicate in Turkish, had a personal cell phone, could read text messages or were illiterate and had a relative to help them at home after discharge were included in the study.

Exclusion Criteria:

* Patients did not volunteered to participate in the study and had not a personal cell phone were excluded in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
postoperative level of anxiety after cataract surgery | 24 months
  The primary point of the study was defined as determining the effect of using SMS, reminding about the intake of medication, on reducing postoperative level of anxiety.

SECONDARY OUTCOMES:
Level of patient satisfaction about received message after cataract surgery | 24 months
  The second point of the study was defined as determining the effect of using SMS, reminding about the intake of medication, on level of patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Dığın, PhD, Principal Investigator — Kırklareli University, Kırklareli, Turkey
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.